CLINICAL TRIAL: NCT01718249
Title: Study of Conscious Behavior Under Low-frequency Deep Brain Stimulation in Chronic and Severe Post-coma Disorders of Consciousness
Acronym: Post-coma DBS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Fondation de l'Avenir (Other); Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: CHU-0126; 2011-A00300-41
Record Dates: First submitted 2012-10-29; First posted 2012-10-31 (Estimated); Last update posted 2017-11-24 (Actual); Status verified 2017-11

CONDITIONS: Chronic and Severe Post-coma Disorders of Consciousness (Permanent Vegetative State, Minimally Conscious State)
Keywords: Deep Brain Stimulation (DBS); Post-coma; Consciousness; Vegetative state; Minimally conscious state
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome; Persistent Vegetative State

STUDY DESIGN:
Who Masked: Participant

ARMS (1):
- deep brain stimulation (Other)
  Interventions: Other: Implantable neurostimulation system

INTERVENTIONS:
Other: Implantable neurostimulation system

SUMMARY:
Chronic post-coma consciousness impairment is a severe handicap. Preliminary studies suggest that deep brain stimulation of the thalamic-tegmental reticular system could improve consciousness disorders, and facilitate the emergence of conscious behavior. The aim of this protocol is to study the effects of deep brain stimulation on conscious behavior, using a patient-based anatomic mapping for stereotactic surgery, and the Coma Recovery Scale-Revised (CRS-R) as clinical assessment criterion.

DETAILED DESCRIPTION:
Total length of inclusion for a patient: 10 months (2 months before electrodes implantation, 8 months after).

ELIGIBILITY:
Inclusion Criteria:

* Patients stably in Vegetative state or Minimally conscious state, since at least 6 months after cerebrovascular accident and 1 year after traumatic brain injury.

Exclusion Criteria:

* Cerebral death, Locked-In Syndrome, blindness, deafness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2012-04 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
CRS-R scores (Coma Recovery Scale-Revised) | after 2 months and after 7 months

SECONDARY OUTCOMES:
signs of awakening at night | during the 10 months of the study
zerit burden interview | at 1 month and at 10 months

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Jacques LEMAIRE, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France